CLINICAL TRIAL: NCT00434343
Title: A Pilot Feasibility Study of Physical Therapy for the Treatment of Urologic Pelvic Pain Syndromes
Brief Title: Physical Therapy Trial for Pelvic Pain
Acronym: UPPCRN-RCT#1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPPCRN RCT1 - PT; U01DK065209 (NIH)
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome; Chronic Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: Interstitial Cystitis; Painful Bladder Syndrome; Chronic Prostatitis; Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Therapeutic Massage (GTM) (Placebo Comparator): Weekly massages consisting of full body Western massage for 1hour.
  Interventions: Other: Global Therapeutic Massage (GTM)
- Myofascial physical therapy (MPT) (Active Comparator): Connective tissue manipulation to all body wall tissues of the abdominal wall, back, buttocks and thighs that clinically were found to contain connective tissue abnormalities and/or myofascial trigger point release to painful myofascial trigger points
  Interventions: Other: Myofascial physical therapy (MPT)

INTERVENTIONS:
Other: Global Therapeutic Massage (GTM)
  Arms: Global Therapeutic Massage (GTM)
Other: Myofascial physical therapy (MPT) — Connective tissue manipulation to all body wall tissues of the abdominal wall, back, buttocks and thighs that clinically were found to contain connective tissue abnormalities and/or myofascial trigger point release to painful myofascial trigger points
  Arms: Myofascial physical therapy (MPT)

SUMMARY:
The purpose of this study is to determine if a randomized trial of physical therapy for pelvic pain is feasible.

DETAILED DESCRIPTION:
This is a pilot study wherein eligible participants will be randomly assigned to receive either myofascial tissue manipulation or global therapeutic massage. Those receiving myofascial tissue manipulation will have targeted internal and external connective tissue manipulation focusing on the muscles and connective tissues of the pelvic floor, hip girdle, and abdomen. Those receiving global therapeutic massage will have non-specific somatic treatment with full-body Western massage.

ELIGIBILITY:
Inclusion Criteria:

* female and male patients who have failed to respond to previous therapies for interstitial cystitis/painful bladder syndrome
* male patients who have failed to respond to previous therapies for chronic prostatitis/chronic pelvic pain syndrome

Exclusion Criteria:

* neurologic disorder affecting bladder
* bladder cancer, prostate cancer, or urethral cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number consenting to join study out of eligible patients approached | 6 months
  This study will recruit both female and male patients who have failed to respond to previous therapies for either Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS) or male patients who have failed to respond to previous therapies for Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS).
Number of times therapists adhered to prescribed therapeutic protocol | 12 weeks
  For each therapy session therapy records are reviewed to determine whether the therapist followed the therapeutic protocol. Each therapy session is scored as adherent or non-adherent and the number of adherent sessions are recorded per participant

SECONDARY OUTCOMES:
Number of adverse events reported by the participants | 12 weeks
  Number of adverse events reported by the participants
Global response assessment (GRA) Global response assessment | 12 weeks
  The global response assessment consists of the following question: "As compared to when you started the study, how would you rate your overall symptoms now?" 1. markedly worse, 2. moderately worse, 3. slightly worse, 4. the same, 5. slightly improved, 6. moderately improved, 7. markedly improved
Tolerability of treatment measured by number of treatment sessions participants completed | 12 weeks
  Treatment session completion was tracked and used to measure tolerability of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Kusek, PhD, Study Director — National Institute of Diabetes & Digestive & Kidney Diseases/National Institutes of Health; Leroy Nyberg, PhD, MD, Study Director — National Institute of Diabetes & Digestive & Kidney Diseases/National Institutes of Health
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Result] FitzGerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2009 Aug;182(2):570-80. doi: 10.1016/j.juro.2009.04.022. Epub 2009 Jun 17. PMID 19535099
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- [Derived] Fitzgerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2013 Jan;189(1 Suppl):S75-85. doi: 10.1016/j.juro.2012.11.018. PMID 23234638